CLINICAL TRIAL: NCT01098669
Title: The Impact of Secondary Lymphedema After Head and Neck Cancer Treatment on Symptoms, Functional Status, and Quality of Life
Brief Title: Impact of Secondary Lymphedema on Symptoms, Functional Status, and Quality of Life After Treatment in Patients With Head and Neck Cancer
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jie Deng, RN, BSN, MSN, Vanderbilt University
Other Study IDs: CDR0000669342; P30CA068485 (NIH); VU-VICC-HN0-9102
Record Dates: First submitted 2010-04-02; First posted 2010-04-05 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Cancer Survivor; Head and Neck Cancer; Lymphedema
Keywords: cancer survivor; lymphedema; head and neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Lymphedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
RATIONALE: Collecting information about the impact of lymphedema on symptoms, functional status, and quality of life after treatment in patients with head and neck cancer may help doctors learn more about the disease and plan the best treatment.

PURPOSE: This phase I trial is studying the effects of secondary lymphedema on symptoms, functional status, and quality of life after treatment in patients with head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To examine the association of secondary lymphedema, symptoms, functional status, and quality of life after treatment in patients with head and neck cancer.
* To examine the possible factors contributing to the development of secondary lymphedema in these patients.

OUTLINE: Participants undergo a physical and external (e.g., submental area) and internal (e.g., larynx, pharynx, and oral cavity) lymphedema examination. Demographics, background, and lymphedema treatment information are also collected. Participants' medical records with head and neck cancer information and treatment are reviewed.

Participants complete surveys on Vanderbilt Head and Neck Symptom (VHNSS), Lymphedema Symptom Intensity and Distress Survey Head and Neck (LSIDS-HN), Functional Assessment Cancer Therapy-Head Neck (FACT-HN), Quality of Life Scale, Hospital Anxiety and Depression Scale (HADS), and Body Image Scale.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosed with head and neck cancer
* At least 3 months since completion of head and neck cancer treatment
* Participating in the Pain and Symptom Management Program at the Vanderbilt-Ingram Cancer Center
* No current evidence of cancer
* No metastatic disease

PATIENT CHARACTERISTICS:

* No other active cancer
* Able to understand informed consent

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No concurrent chemotherapy or radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult head and neck cancer survivors
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2009-12; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Association between the severity of lymphedema with symptoms, functional status, and quality of life | Cross-sectional
Factors contributing to the development of secondary lymphedema | Cross-sectional Study

CONTACTS AND LOCATIONS:
Overall Officials: Jie Deng, RN, BSN, MSN, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (2):
- United States (2):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee